CLINICAL TRIAL: NCT05138484
Title: Clinical Evaluation of a Mouthwash Containing Malva Sylvestris Extract and Its Role in Reducing Oral Biofilm and Gingival Inflammation. A Randomized, Triple Masked Clinical Trial.
Brief Title: Clinical Evaluation of a Mouthwash Containing Malva Sylvestris Extract.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aravena, Pedro, DDS, PhD (Other)
Collaborators: Universidad Austral de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ORD 181
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2019-05

CONDITIONS: Periodontal Diseases
Keywords: Periodontal diseases; Inflammation; Malva sylvestris; Mouthwashes
MeSH Terms: conditions — Periodontal Diseases; Inflammation | interventions — chlorhexidine gluconate

STUDY DESIGN:
Intervention Model Description: Two examiners recorded the data: sex, age, hygiene habits, systemic diseases, use of drugs and smoking.
  Clinical examination and registration of clinical indexes: Basic Periodontal Examination, Gingival Bleeding Index, Bacterial plaque index.
  Another investigator performed, through simple randomization, the patient's assignment to one of the three parallel study groups:
  G.1 (Positive control 0.12% chlorhexidine digluconate) G.2 (Negative control vehicle mouthwash) G.3 (experimental group 10% mouthwash of M. sylvestris extract). To each patient was delivering a 150 ml bottle with the corresponding mouthwash. The indications for posology were: rinse with 10 ml of mouthwash for 1 minute in the mouth, every 12 hours for 7 days. To the follow-up of the intervention, was made telephone calls at least once a day to remember the rinse.
  The re-evaluation was performed 7 days after the first appointment.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Each clinical record was coded by number, group and each group was assigned a color, which was stamped on the bottle of each mouthwash (bottles were of the same appearance).
  The masking mechanisms through coding by number, group and color, ensured that the patients did not know the specific mouthwash they received; examiners E.A and A.N were limited only to assessing the clinical aspects; and the data analysis was performed with the database using numerical coding. Only researcher B.B was aware of the real assignment by color, with its corresponding study group and number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- M. sylvestris mouthwash (Experimental): using 10 ml, rinse for one minute, 1 time every 12 hours for 7 days.
  Interventions: Drug: experimental group 10% mouthwash of M. sylvestris extract
- CHX mouthwash (Active Comparator): using 10 ml, rinse for one minute, 1 time every 12 hours for 7 days.
  Interventions: Drug: experimental group 10% mouthwash of M. sylvestris extract
- Placebo mouthwash (Placebo Comparator): using 10 ml, rinse for one minute, 1 time every 12 hours for 7 days.
  Interventions: Drug: experimental group 10% mouthwash of M. sylvestris extract

INTERVENTIONS:
Drug: experimental group 10% mouthwash of M. sylvestris extract — To each patient was delivering a 150 ml bottle with the corresponding mouthwash. The indications for posology were: rinse with 10 ml of mouthwash for 1 minute in the mouth, every 12 hours for 7 days. To the follow-up of the intervention, was made telephone calls at least once a day to remember the rinse.
  Other Names: Positive control 0.12% chlorhexidine digluconate; Negative control vehicle mouthwash

SUMMARY:
Background: For centuries, plants (and / or their products) were the only resource available for the prevention and treatment of many diseases. However, its indiscriminate use without phytochemical, pharmacological and toxicological knowledge is a concern for health. The Malva sylvestris (family Malvaceae and popularly known as Malva) is mentioned in the literature as an ethnopharmacological medicine with anti-inflammatory, antimicrobial, wound healing and other properties. For this reason, M. sylvestris presents empirical indications in dentistry, mainly in the treatment of periodontal diseases (gingivitis and periodontitis), which are highly prevalent worldwide. However, scientific evidence is scarce in information that supports the biological properties and clinical benefits attributed to it.

Objective: The objective of this study was to evaluate the effect of a mouthwash based on Malva sylvestris in the control of gingival inflammation and dental biofilm.

Methods: A randomized, three-group, triple-masked clinical trial was designed. Patients from the Center of Dental Clinics of the Austral University of Chile participated with a diagnosis of gingivitis and chronic periodontitis. They were distributed randomly in three study groups: 1. Chlorhexidine mouthwash 0.12%; 2. Mouthwash with extract of M. sylvestris and 3. Mouthwash control group. The indications and dosage were identical for all groups: rinse with 10 ml, for 1 minute, every 12 hours for 7 days. The gingival index and plaque control record were recorded at the beginning and end of the follow-up period (7 days). The results obtained between the groups were compared through normality test and group analysis (ANOVA/Mann-Whitney/Dunnet p <0.05).

Results: The pharmacological potential of M. sylvestris was determined in the reduction of the plaque control record and gingival index.

DETAILED DESCRIPTION:
Design:

It´s designed a randomized clinical trial of three parallel groups, triple masking. The study and informed consent document were reviewed and approved by the Comité Ético Científico of Servicio de Salud Valdivia (ORD 181/2017) and written according to the CONSORT (EQUATOR Network) writing guidelines.

Population:

The participants were selected from the Department of Oral and Periodontal Surgery of the Dental Clinic Center of the Universidad Austral de Chile (UACh) (Valdivia, southern Chile) during the months of October 2017 to December 2018.

Sample size:

For the calculation of the sample size, the effectiveness of the use of CHX mouthwash was considered over placebo, a standardized mean in the reduction of the gingival index according to Loe & Silness (1963) parameters of 0.21 (95% CI: 0.1-0.31) (15). Probability of error of 5%, statistical power of 80% and margin of loss of follow-up or absence of data of 20%. The participation of 18 subjects was determined by study group (calculation algorithm: "power two means 1.21 1, sd1 (0.2) sd2 (0.2) knowns", STATA V.14.0, STATASp, Texas, USA).

Preparation of M. sylvestris extract and mouthwash:

For the preparation of the mouthwash of M. sylvestris, the leaves registered in the herbarium of the University of Sao Paulo (USP) were used. Identification number ESA voucher # 121403. The leaves were dried in a forced circulation oven for 24 h, at 40 °C, and then crushed. The extraction was carried out with absolute ethanol under climatic control (25 °C) and subjected to exhaustive extraction (7 days) in a rotating shaker protected against light. In the extraction sequence, the samples were filtered, concentrated by evaporation and lyophilized for 72 h. The EEM was stored at -20 °C. The chemical monitoring was conducted by HPLC MS/MS technique (33). The mouthwash based on M. sylvestris was prepared at a standard concentration of 10% using a 1% ethanol vehicle for preservation of compounds at a concentration compatible with morphofunctional stability (32,33). The control mouthwash presents the same vehicle and composition as the previous one but is exempted from the active compound and the CHX mouthwash was prepared at a concentration of 0.12% with the same vehicle as an accentuated at a concentration of 0.12%.

Periodontal indices record:

Prior to the clinical trial, two examiners (E.A and A.N) underwent a calibration process for the registration of clinical indices (BPE, gingival index and plaque control record) with a specialist in periodontics. To this end, 10 patients from the Center of Dental Clinics of the UACh were evaluated, diagnosed by the specialist with gingival index (GI) over 90% and moderate chronic periodontitis in one of their dental sextants. Inter-examiner and intra-examiner kappa index of 0.89 and 0.80, respectively.

The objective and methodology of the study were explained to the patients who fulfilled the selection criteria and who had already been previously diagnosed. Those who agreed to participate, signed an informed consent document.

On the day of the appointment, the examiners, confirmed the fulfillment of the selection criteria and recorded the data: sex, age, hygiene habits, systemic diseases, use of drugs and smoking.

Then we proceeded to the clinical examination and the following indices were evaluated:

* Basic Periodontal Examination (BPE): The mouth is divided into sextants and using a WHO-standardized periodontal probe, the probing of each tooth is performed in 3 points (mesial, medial and distal) by vestibular and lingual-palatal of each tooth, registering the highest value per sextant, according to the following coding: 0 (healthy tissue), 1 (positive bleeding, absence of periodontal pocket), 2 (presence of tartar, defective fillings, black area of the probe completely visible), 3 (periodontal pocket greater than 5.5 mm) (35).
* Gingival Index (GI): With a WHO-standardized periodontal probe, the buccal, lingual and interdental papillae marginal gingival are probed, using a four-point scale from 0 (absence of inflammation) to 3 (severe inflammation) (37,38).
* Plaque control record (PC): 5 drops of Plaque Revealing Solution are applied, and the patient is instructed to make movements with the tongue in such a way that it touches all dental surfaces in a time of 15 seconds. The vestibular, lingual and interproximal surfaces of all the teeth are then examined. To calculate the index, add the total number of dental surfaces with plaque, divide this number by the total number of surfaces present in the mouth and multiply by 100 (39).

Randomization and use of mouthwash:

The randomization and masked identification of the mouthwashes was done by a single researcher (B.B.). All mouthwashes were dispensed in a 150 mL white vial and each content was identified by a different colored marker known only to the investigator in charge.

To determine the randomization of each patient within the three groups, the page www.random.org was used, with the numbers 1,2 or 3 corresponding to the groups G1, G2 and G3, respectively, being returned as a result.

For this, the patients were randomized into 3 parallel study groups:

* G1 (Green): Positive Control (0.12% CHX)
* G2 (Orange): Negative control (alcohol vehicle mouthwash 0.1%)
* G3 (Yellow): Experimental group (10% mouthwash of M. sylvestris extract). After the clinical examination, another researcher (V.Ll.) recorded in each clinical record the patient's coding assigned by number, group and color. He delivered the bottle and posology to each patient corresponding to the randomized group, having to rinse with 10 ml of mouthwash for 1 minute in the mouth, every 12 h for 7 days. To confirm the follow-up of the intervention, the same researcher made telephone calls at least once a day to remember the daily rinse. The instructions were delivered verbally and in writing.

The re-evaluation of the patients was carried out 7 days after the first appointment, by the same examiner registering the PBE, GI and PC indices.

Control of risk of bias:

The masking mechanisms through coding by number, group and color, ensured that the patients did not know the specific mouthwash they received; examiners E.A and A.N were limited only to assessing clinical aspects and data analysis was performed with the database using numerical coding. Only researcher B.B was aware of the real assignment by color, with its corresponding study group and number.

To control the risk of random bias in the changes of hygiene habits of the participants on the registration of the periodontal indices, the frequency of brushing, type of toothpaste and use of oral antiseptic mouthwashes was registered; indicating to each participant to maintain these habits without needing to change the oral hygiene frequency.

Statistics:

Mouthwash study groups were defined as an independent variable. The PC and GI analyzed at the beginning and 7 days after the intervention of the study were defined as dependent variable. An analysis of descriptive statistics of the following data was performed: sex (male/female), age (in years), frequency of brushing/day, smoking (smokes over 10 cigarettes/day), presence of chronic disease (Yes/No) and medication consumption (Yes/No). In addition, the values of PC and GI. The continuous variables were presented as average values (Standard Deviation - SD).

In the analytical statistics, the normality of the data was analyzed by the Shapiro Wilk test (p> 0.05). To compare the indices between the 3 groups before and after the intervention, the data were analyzed by repeated measures ANOVA (MR). The nonparametric data were presented as scatter plot of the samples, comparison with T-test to detect differences.

Considering the variability of the initial data of the patients belonging to each study group that can generate a result bias, an analysis of covariance (ANCOVA) of the baseline data was performed. To check the study hypotheses, the mean values were compared, with a 95% confidence interval of the results between study groups, establishing a level of significance of p <0.05

ELIGIBILITY:
Inclusion Criteria:

* Code equal of higher than 2 (Basic Periodontal Examination-BPE).
* I or II ASA classification.
* Without periodontal treatment on past three months.

Exclusion Criteria:

* Acute infection
* Dental trauma
* Alveolar osteitis (Dry socket)
* Elderly dependent patients
* Orthodontic appliances
* Antibiotic therapy
* Analgesic therapy
* Heavy smokers
* Menstrual period
* Pregnants
* Lactating woman

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Basic periodontal examination | 7 days
  The mouth is divided into sextants and using a WHO-standardized periodontal probe (Hu-FriedyⓇ), the probing of each tooth is performed in 3 points (mesial, medial and distal) by vestibular and lingual -palatal of each tooth, registering the highest value per sextant, according to the following coding: 0 (healthy tissue), 1 (positive bleeding, absence of periodontal pocket), 2 (presence of tartar, defective fillings, black area of the probe completely visible), 3 (black area of the probe partially visible, periodontal pocket of 3.5 - 5.5 mm), 4 (black area of the probe below the gingival margin, periodontal pocket greater than 5.5 mm).
Gingival index | 7 days
  With a WHO-standardized periodontal probe (Hu-FriedyⓇ), the buccal, lingual and interdental papillae marginal gingivae are probed, using a four-point scale from 0 (absence of inflammation) to 3 (severe inflammation)
Plaque control record | 7 days
  5 drops of Bacterial Plaque Revealing Solution (Caristop-Revelador DUAL TONE, MAVERⓇ) are applied and the patient is instructed to make movements with the tongue in such a way that it touches all dental surfaces in a time of 15 seconds . The vestibular, lingual and interproximal surfaces of all the teeth are then examined. To calculate the index, add the total number of dental surfaces with bacterial plaque, divide this number by the total number of surfaces present in the mouth and multiply by 100

CONTACTS AND LOCATIONS:
Overall Officials: Bruna Benso, PhD, Principal Investigator — Faculty of Medicine, Pontificia Universidad Católica de Chile
Locations (1):
- Universidad Austral de Chile, Valdivia, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pihlstrom BL, Michalowicz BS, Johnson NW. Periodontal diseases. Lancet. 2005 Nov 19;366(9499):1809-20. doi: 10.1016/S0140-6736(05)67728-8. PMID 16298220
- [Background] Hooks KB, O'Malley MA. Dysbiosis and Its Discontents. mBio. 2017 Oct 10;8(5):e01492-17. doi: 10.1128/mBio.01492-17. PMID 29018121
- [Background] Gao L, Xu T, Huang G, Jiang S, Gu Y, Chen F. Oral microbiomes: more and more importance in oral cavity and whole body. Protein Cell. 2018 May;9(5):488-500. doi: 10.1007/s13238-018-0548-1. Epub 2018 May 7. PMID 29736705
- [Background] Murakami S, Mealey BL, Mariotti A, Chapple ILC. Dental plaque-induced gingival conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S17-S27. doi: 10.1111/jcpe.12937. PMID 29926503
- [Background] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Clin Periodontol. 2018 Jun;45 Suppl 20:S149-S161. doi: 10.1111/jcpe.12945. PMID 29926495
- [Background] Rafiei M, Kiani F, Sayehmiri F, Sayehmiri K, Sheikhi A, Zamanian Azodi M. Study of Porphyromonas gingivalis in periodontal diseases: A systematic review and meta-analysis. Med J Islam Repub Iran. 2017 Sep 12;31:62. doi: 10.18869/mjiri.31.62. eCollection 2017. PMID 29445691
- [Background] Hajishengallis G. Periodontitis: from microbial immune subversion to systemic inflammation. Nat Rev Immunol. 2015 Jan;15(1):30-44. doi: 10.1038/nri3785. PMID 25534621
- [Background] Topcuoglu N, Kulekci G. 16S rRNA based microarray analysis of ten periodontal bacteria in patients with different forms of periodontitis. Anaerobe. 2015 Oct;35(Pt A):35-40. doi: 10.1016/j.anaerobe.2015.01.011. Epub 2015 Jan 29. PMID 25638399
- [Background] Teles RP, Teles FR. Antimicrobial agents used in the control of periodontal biofilms: effective adjuncts to mechanical plaque control? Braz Oral Res. 2009;23 Suppl 1:39-48. doi: 10.1590/s1806-83242009000500007. PMID 19838557
- [Background] Larsen T, Fiehn NE. Dental biofilm infections - an update. APMIS. 2017 Apr;125(4):376-384. doi: 10.1111/apm.12688. PMID 28407420
- [Background] Loe H, Schiott CR, Karring G, Karring T. Two years oral use of chlorhexidine in man. I. General design and clinical effects. J Periodontal Res. 1976 Jun;11(3):135-44. doi: 10.1111/j.1600-0765.1976.tb00061.x. No abstract available. PMID 133217
- [Background] Gunsolley JC. Clinical efficacy of antimicrobial mouthrinses. J Dent. 2010 Jun;38 Suppl 1:S6-10. doi: 10.1016/S0300-5712(10)70004-X. PMID 20621242
- [Background] Collins JR, Olsen J, Cuesta A, Silva-Vetri M, Hernandez M, Romanos G, Rajendra Santosh AB, Palma P. In vitro microbiological analysis on antibacterial, anti-inflammatory, and inhibitory action on matrix metalloproteinases-8 of commercially available chlorhexidine digluconate mouth rinses. Indian J Dent Res. 2018 Nov-Dec;29(6):799-807. doi: 10.4103/ijdr.IJDR_406_17. PMID 30589011
- [Background] James P, Worthington HV, Parnell C, Harding M, Lamont T, Cheung A, Whelton H, Riley P. Chlorhexidine mouthrinse as an adjunctive treatment for gingival health. Cochrane Database Syst Rev. 2017 Mar 31;3(3):CD008676. doi: 10.1002/14651858.CD008676.pub2. PMID 28362061
- [Background] Gurgan CA, Zaim E, Bakirsoy I, Soykan E. Short-term side effects of 0.2% alcohol-free chlorhexidine mouthrinse used as an adjunct to non-surgical periodontal treatment: a double-blind clinical study. J Periodontol. 2006 Mar;77(3):370-84. doi: 10.1902/jop.2006.050141. PMID 16512751
- [Background] Van Strydonck DA, Slot DE, Van der Velden U, Van der Weijden F. Effect of a chlorhexidine mouthrinse on plaque, gingival inflammation and staining in gingivitis patients: a systematic review. J Clin Periodontol. 2012 Nov;39(11):1042-55. doi: 10.1111/j.1600-051X.2012.01883.x. Epub 2012 Sep 7. PMID 22957711
- [Background] Baker K. Mouthrinses in the prevention and treatment of periodontal disease. Curr Opin Periodontol. 1993:89-96. PMID 8401852
- [Background] Tartaglia GM, Kumar S, Fornari CD, Corti E, Connelly ST. Mouthwashes in the 21st century: a narrative review about active molecules and effectiveness on the periodontal outcomes. Expert Opin Drug Deliv. 2017 Aug;14(8):973-982. doi: 10.1080/17425247.2017.1260118. Epub 2016 Nov 20. PMID 27835926
- [Background] Newman DJ, Cragg GM. Natural Products as Sources of New Drugs from 1981 to 2014. J Nat Prod. 2016 Mar 25;79(3):629-61. doi: 10.1021/acs.jnatprod.5b01055. Epub 2016 Feb 7. PMID 26852623
- [Background] Lazar V, Saviuc CM, Chifiriuc MC. Periodontitis and Periodontal Disease - Innovative Strategies for Reversing the Chronic Infectious and Inflammatory Condition by Natural Products. Curr Pharm Des. 2016;22(2):230-7. doi: 10.2174/138161282202151221124307. PMID 26561076
- [Background] Araujo MWB, Charles CA, Weinstein RB, McGuire JA, Parikh-Das AM, Du Q, Zhang J, Berlin JA, Gunsolley JC. Meta-analysis of the effect of an essential oil-containing mouthrinse on gingivitis and plaque. J Am Dent Assoc. 2015 Aug;146(8):610-622. doi: 10.1016/j.adaj.2015.02.011. PMID 26227646
- [Background] Freires IA, Denny C, Benso B, de Alencar SM, Rosalen PL. Antibacterial Activity of Essential Oils and Their Isolated Constituents against Cariogenic Bacteria: A Systematic Review. Molecules. 2015 Apr 22;20(4):7329-58. doi: 10.3390/molecules20047329. PMID 25911964
- [Background] Van Leeuwen MP, Slot DE, Van der Weijden GA. Essential oils compared to chlorhexidine with respect to plaque and parameters of gingival inflammation: a systematic review. J Periodontol. 2011 Feb;82(2):174-94. doi: 10.1902/jop.2010.100266. Epub 2010 Nov 2. PMID 21043801
- [Background] Barros L, Carvalho AM, Ferreira IC. Leaves, flowers, immature fruits and leafy flowered stems of Malva sylvestris: a comparative study of the nutraceutical potential and composition. Food Chem Toxicol. 2010 Jun;48(6):1466-72. doi: 10.1016/j.fct.2010.03.012. Epub 2010 Mar 15. PMID 20233600
- [Background] Gasparetto JC, Martins CA, Hayashi SS, Otuky MF, Pontarolo R. Ethnobotanical and scientific aspects of Malva sylvestris L.: a millennial herbal medicine. J Pharm Pharmacol. 2012 Feb;64(2):172-89. doi: 10.1111/j.2042-7158.2011.01383.x. Epub 2011 Nov 4. PMID 22221093
- [Background] Razavi SM, Zarrini G, Molavi G, Ghasemi G. Bioactivity of malva sylvestris L., a medicinal plant from iran. Iran J Basic Med Sci. 2011 Nov;14(6):574-9. PMID 23493458
- [Background] Guarrera PM. Traditional phytotherapy in Central Italy (Marche, Abruzzo, and Latium). Fitoterapia. 2005 Jan;76(1):1-25. doi: 10.1016/j.fitote.2004.09.006. PMID 15664457
- [Background] DellaGreca M, Cutillo F, D'Abrosca B, Fiorentino A, Pacifico S, Zarrelli A. Antioxidant and radical scavenging properties of Malva sylvestris. Nat Prod Commun. 2009 Jul;4(7):893-6. PMID 19731587
- [Background] Benso B, Rosalen PL, Alencar SM, Murata RM. Malva sylvestris Inhibits Inflammatory Response in Oral Human Cells. An In Vitro Infection Model. PLoS One. 2015 Oct 19;10(10):e0140331. doi: 10.1371/journal.pone.0140331. eCollection 2015. PMID 26479870
- [Background] Benso B, Franchin M, Massarioli AP, Paschoal JA, Alencar SM, Franco GC, Rosalen PL. Anti-Inflammatory, Anti-Osteoclastogenic and Antioxidant Effects of Malva sylvestris Extract and Fractions: In Vitro and In Vivo Studies. PLoS One. 2016 Sep 19;11(9):e0162728. doi: 10.1371/journal.pone.0162728. eCollection 2016. PMID 27643502
- [Background] Offenbacher S, Barros SP, Beck JD. Rethinking periodontal inflammation. J Periodontol. 2008 Aug;79(8 Suppl):1577-84. doi: 10.1902/jop.2008.080220. PMID 18673013
- [Background] Jeffcoat MK, McGuire M, Newman MG. Evidence-based periodontal treatment. Highlights from the 1996 World Workshop in Periodontics. J Am Dent Assoc. 1997 Jun;128(6):713-24. doi: 10.14219/jada.archive.1997.0294. PMID 9188228
- [Background] DRIPPS RD, LAMONT A, ECKENHOFF JE. The role of anesthesia in surgical mortality. JAMA. 1961 Oct 21;178:261-6. doi: 10.1001/jama.1961.03040420001001. No abstract available. PMID 13887881
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Background] Ainamo J, Bay I. Problems and proposals for recording gingivitis and plaque. Int Dent J. 1975 Dec;25(4):229-35. PMID 1058834
- [Background] O'Leary TJ, Drake RB, Naylor JE. The plaque control record. J Periodontol. 1972 Jan;43(1):38. doi: 10.1902/jop.1972.43.1.38. No abstract available. PMID 4500182